CLINICAL TRIAL: NCT00247481
Title: A Multicentre, Randomised, Double-Blind, Non-Comparative Phase II Trial Of ZD1839 (Iressa™) And Placebo In Combination With Chemotherapy With Docetaxel As First-Line Treatment In Patients With Metastatic Breast Cancer
Brief Title: ZD1839 (Iressa™) In Combination With Docetaxel As First-Line Treatment In Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D7913C00148; 1839IL/0148
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib; Docetaxel

INTERVENTIONS:
Drug: Gefitinib
Drug: Docetaxel

SUMMARY:
This is a multicentre, randomised (2:1), double blind, non-comparative phase II trial of ZD1839 and placebo in combination with chemotherapy in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer at a metastatic stage.
* Uni- or bi-dimensionally measurable lesions (10 mm or 20 mm) according to the Response Evaluation Criteria in Solid Tumours (RECIST) criteria
* World Health Organisation (WHO) performance status (PS) of 0 to 2
* Life expectancy of greater than 12 weeks
* Normal cardiac function (left ventricular ejection fraction [LVEF] by isotopic examination greater than or equal to 55%)

Exclusion Criteria:

* Symptomatic lepto-meningeal metastasis
* Concomitant infectious disease
* Any unresolved chronic toxicity greater than CTC grade 2 from previous anticancer therapy
* Incomplete healing from previous oncologic or other surgery
* Absolute neutrophil count (ANC) less than 1.5 x 109/litre (L) or platelets less than 100 x 109/L
* Serum creatinine greater than 1.5 times the ULRR or clearance < 60 ml/min
* ALT or AST greater than 2.5 times the ULRR
* ALP > 5 times the ULRR
* ALP > 2.5 times the ULRR and ALT or AST greater than 1.5 times the ULRR

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77
Dates: Start 2002-09; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
To estimate the overall response rates (complete response [CR] and partial response [PR]) in the ZD1839-treated group and the placebo-treated group.

SECONDARY OUTCOMES:
o To assess progression-free survival (PFS) in the ZD1839-treated group and the placebo-treated group.
o To estimate the duration of response in the ZD1839-treated group and the placebo treated group
o To estimate overall survival in the ZD1839-treated group and the placebo-treated group
o To estimate time to treatment failure (TTF) in the ZD1839-treated group and the placebo treated group

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, MD, Study Director — AstraZeneca
Locations (5):
- France (5):
  - Research Site, Dijon
  - Research Site, Paris
  - Research Site, Saint-Cloud
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Villejuif